CLINICAL TRIAL: NCT06400732
Title: Post Market Evaluation of Clinical Safety and Performance of the Fitbone Transport and Lengthening System
Status: Active, not recruiting | Type: Observational
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-FBBT-23
Record Dates: First submitted 2024-04-29; First posted 2024-05-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Fractures, Bone; Fractures, Closed; Fractures, Open; Fracture of Femur; Fracture Nonunion; Fracture of Tibia; Limb Deformity; Limb Fracture; Limb Defect; Limb Asymmetry
Keywords: Limb Lengthening; Limb Deformity Correction; Bone Transport
MeSH Terms: conditions — Fractures, Bone; Fractures, Closed; Fractures, Open; Femoral Fractures; Fractures, Ununited; Tibial Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: Participants treated for a limb defect with the Fitbone Transport and Lengthening System
  Interventions: Device: Fitbone Transport and Lengthening System

INTERVENTIONS:
Device: Fitbone Transport and Lengthening System — Implantation of the intramedullary Fitbone Transport Nail and subsequent bone segment transport and, optionally, lengthening.
  Other Names: Fitbone Transport Nail

SUMMARY:
This is an open-label, prospective, observational, post-market, uncontrolled, multi-center study intended to evaluate the safety and clinical performance of the FITBONE Transport and Lengthening Nail when used according to the manufacturer's Instructions for Use. The FITBONE Transport & Lengthening Nail is a variant of the FITBONE TAA Nail, which has been commercially available in the US since 2017. The clinical performance and safety of the medical device have been assessed based on mechanical and biomechanical tests and clinical data obtained from scientific publications on equivalent products. This study intends to prospectively obtain clinical safety and performance data on the device, as used according to the manufacturer's Instructions for Use, in the real-world clinical setting.

The data obtained from this study will also be used to provide additional clinical evidence to support product registrations, as required by various regulatory bodies outside the US.

Eligible participants will have been selected by their physician to be treated with the FITBONE Transport and Lengthening System as part of treatment for their condition or injury. All procedures will be according to the physician's standard care practices. There are no study-specific procedures or requirements for participants in this study.

DETAILED DESCRIPTION:
This prospective, observational clinical study intends to actively collect clinical data related to the use of the FITBONE Transport and Lengthening System in a representative number of users and patients, observed in the short (<1yr) and medium (approximately 1 and 2 years) term after implantation of the device.

Co-Primary Endpoints:

Primary Safety Endpoint: Percentage of unplanned reoperation and/or revision surgery. Instances of re-operation and/or revision as categorized as "planned" or "unplanned" by the surgeon.

Primary Performance Endpoint: Percentage of achievement of planned length. Length of the planned transport (and lengthening when applicable) vs the actual overall length of the segment at the time of nail extraction.

Secondary Endpoints:

* Bone Healing: Radiographic evidence of healing of 3 out of 4 cortices
* Consolidation Index: Time to achieve bone healing (days)/ achieved length (cm)
* Distraction Index: Time of distraction (days)/ achieved length (cm)
* Nail Reliability: Ratio between the number of successfully completed lengthening treatments and the number of implanted lengthening devices
* Nail Accuracy: Ratio between the achieved length and the planned length
* Time to achieve transport and lengthening
* Loss of Range of Motion at full consolidation: degrees from baseline
* Nail Extraction complications/failures
* Patient-reported outcome measures
* Mobility measures
* Adverse events

Safety Endpoint:

The percentage of cases in which unplanned reoperations and/or revision surgery occurred.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Expressed willingness to participate in the study by signing and dating the informed consent form
3. Has a segmental bone defect, or limb length defect of at least 2 mm up to ≤ 120 mm, considered suitable for correction with an intramedullary lengthening nail, as confirmed by radiographs.

Exclusion Criteria:

1. Conditions that tend to retard healing such as blood supply limitations, peripheral vascular disease, or evidence of inadequate vascularity
2. Poor bone quality that would prevent adequate fixation of the device
3. Compromised capacity for healing
4. Metal allergies and sensitivities
5. Patients in which the implant would cross open, healthy epiphyseal growth plates
6. Insufficient intramedullary space which would lead to cortical weakening or vascular damage during implantation
7. Body weight of > 100 kg
8. No free access for proximal insertion of the intramedullary transport and lengthening nail (e.g., coxa valga)
9. No reliable exclusion of bone infection
10. Expected non-compliance, mentally ill patient or patient with clouded consciousness
11. Pregnancy
12. Pre-existing nerve palsies
13. Bone defect larger than 120 mm
14. Gustilo Open Fracture Classification Grade IIIB or IIIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are indicated, as described in the Instructions for Use, for treatment with the Fitbone Transport and Lengthening System for correction of limb deformity.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety - Percentage of unplanned reoperation and/or revision surgery. | 1 year post-operative
  Instances of re-operation and/or revision as categorized as "planned" or "unplanned" by the surgeon. Specifically, adverse events consisting of re-operation/revision surgery deemed to be related to the device or procedure will be tabulated and the incidence will be determined by dividing this by the total number of patients treated (expressed as %).
Performance - Percentage of achievement of planned lengthening. Length of the planned transport (and lengthening when applicable) vs the actual overall length of the segment at the time of nail extraction. | 1 year post-operative
  Incidence of participants in which successful attainment of target lengthening/distraction was obtained. Specifically, the outcome measure will be based on the difference between the physician's pre-specified target length/distraction to be obtained and the actual lengthening/distraction obtained following treatment. The physician will make a determination if this difference is acceptable for each subject. The incidence of successful lengthening will be determined by the number of clinical acceptable results divided by the total number of patients treated (expressed as %).

SECONDARY OUTCOMES:
Effectiveness - Bone Healing | 1 year and 2 years post-operative
  Radiographic evidence of healing of 3 out of 4 cortices
Effectiveness - Consolidation Index | 1 year and 2 years post-operative
  Time to achieve bone healing (days)/ achieved length (cm)
Effectiveness - Distraction Index | 1 year post-operative
  Time of distraction (days)/ achieved length (cm)
Effectiveness - Nail Reliability | 1 year post-operative
  Ratio between the achieved length and the planned length
Effectiveness -Time to Transport and Lengthening | 1 year post-operative
  Time to achieve transport and lengthening
Effectiveness - Range of Motion | 1 year and 2 years post-operative
  Loss of Range of Motion at full consolidation; degrees from baseline
Safety -Nail Extraction | 1 year post-operative
  Nail extraction complications/failures
Effectiveness - Patient Reported Outcome Measures (PROMs) | 1 year and 2 years post-operative
  Improvement in PROMS scores (Pain, Quality of Life) obtained per standard of care
Effectiveness - Mobility Measures | approximately 2 years post-operative
  Improvement in gait analysis
Safety - Adverse Events | Index surgery through study completion; approximately 2 years post-operative
  Evaluation and classification of all adverse events including device-related, procedure-related and serious adverse events.

OTHER OUTCOMES:
Primary Safety Endpoint | 1 year and 2 years post-operative
  The percentage of cases in which unplanned reoperations and/or revision surgery occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Erturan, MD, JD, Study Director — Orthofix Inc.
Locations (9):
- United States (9):
  - Cedars Sanai Medical Center, Los Angeles, California
  - University California - Irvine, Orange, California
  - Emory University School of Medicine / Grady Memorial Hospital, Atlanta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - The Research Foundation for SUNY, Buffalo, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Virginia Health, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No